CLINICAL TRIAL: NCT04717271
Title: Effects of Kinesthetic Stimuli Provided by the Physiotherapist During XBOX Kinect Training on the Functionality of People With Parkinson's Disease: A Blind Randomized Clinical Trail
Brief Title: Effects of Kinesthetic Stimuli During XBOX Kinect Training on People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pâmela
Record Dates: First submitted 2021-01-04; First posted 2021-01-22 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Physical Therapy Specialty; Virtual Reality; International Classification of Functioning; Disability and Health; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A single-blind, parallel-group and randomized clinical trial
Who Masked: Investigator
Masking Description: A experient physical therapy will be responsible for assessments of all participants without knowing the group allocation of which.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement Guidance Group (MVG) (Experimental): In the MVG Group, the physiotherapist will provide kinesthetic stimuli by assisting manually the participant movements.
  Interventions: Other: Movement Guidance Group
- No Movement Guidance Group (NO-MVG) (Experimental): In the NO-MVG, the involvement of the physiotherapist will be restricted to guarantee the safety of the participant.
  Interventions: Other: No Movement Guidance Group

INTERVENTIONS:
Other: Movement Guidance Group — Participants of the MVG will received kinesthetic stimuli by manual assistance of the physiotherapist, which has the intention of guiding and improving the quality of movement during XBOX Kinect training for balance and gait.
  Each session consisted of 10 minutes of warm-up and 40 minutes of XBOX Kinect training, using 4 different exergames.
  Other Names: MVG
  Arms: Movement Guidance Group (MVG)
Other: No Movement Guidance Group — Participants of the NO-MVG will not received kinesthetic stimuli by manual assistance of the physiotherapist during XBOX Kinect training for balance and gait.
  They will perform the exercises without any manual correction. Although, the physiotherapist will be present during all session to ensure their safety.
  Each session consisted of 10 minutes of warm-up and 40 minutes of XBOX Kinect training, using 4 different exergames.
  Other Names: NO-MVG
  Arms: No Movement Guidance Group (NO-MVG)

SUMMARY:
A single-blind, parallel-group, randomised trial will be conducted in Sao Paulo, Brazil. People with Parkinson's Disease (PD) will be recruited at "Brazil Parkinson Association" (BPA), a non-governmental association of PD care, and randomly allocated in two groups: the Movement Guidance Group (MVG) and NO-MVG Group. Both groups will perform XBOX Kinect training for balance and gait. However, the MVG will receive kinesthetic stimuli manually by the physiotherapist (PT) to improve the participant movements while the NO-MVG Group will not, the presence of the PT will be restrict to only guarantee the participant safety.

DETAILED DESCRIPTION:
BACKGROUND: Despite evidences indicate the benefit of motor interventions based on video games in people with Parkinson's Disease (PD), practice guidelines for the therapeutic use in physiotherapy were still not established. Although visual and auditory stimuli provided by video games are pointed as one of the main advantages for their therapeutic use, the effects of kinesthetic stimuli offered through physical therapist manual intervention during this type of training in people with PD have not been investigated yet. The answer to this question is relevant to guide the physical therapist (PT) conduct during this kind of intervention.

PURPOSE: To compare the effects of motor training using video games with and without kinesthetic stimuli offered by physical therapist manual guidance during intervention on the functionality of people with PD.

METHODS: A blind randomized clinical trial in people with idiopathic PD, staging of 1 to 3 according to disability scale of Hoehn and Yahr, will be performed. Participants will be randomized into two groups: the Movement Guidance Group (MVG) and NO-MVG Group. Both groups will receive 8 individual sessions, twice a week, for 4 weeks. Each session consist of 10 minutes of warm-up and 40 minutes of XBOX Kinect training for balance and gait. In the MVG Group, the PT will provide kinesthetic stimuli by assisting manually the participant movements. In the NO-MVG Group, the involvement of the PT will be restricted to ensure participant safety. The two groups will be evaluated before (BT) and after (AT) training and after 60 days (follow-up). A blind physiotherapist will conduct the assessments. Measurements are categorized according to the International Functioning Classification (ICF), those associated with the activity level were established as primary measures: Balance Evaluation Systems Test (BESTest); International Falls Effectiveness Scale (FES-I); 30-second Gait Test; Six Minute Walk Distance (6MWD); Five Times Sit to Stand Test (FTSTS) and Unified Parkinson's Disease Rate Scale (UPDRS) session II. Secondary measures were the evaluation of function using UPDRS session III; Rapid Turns Test (RTT); Montreal Cognitive Assessment (MOCA); Geriatric Depression Scale (GDS-15), and participation using the Parkinson's Disease Quality of Life Questionnaire (PDQ-39).

STATISTICAL ANALYSIS: An ANOVA to repeated measures will be use, having as factors: group (MVG Group and NO-MVG Group) and evaluations (BT, AT and FU). Followed by post hoc Tukey Test to the significance factors. A significance of 5% will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease diagnosis according to Parkinson's Disease Society Brain Bank of London criteria
* Active treatment with levodopa
* Stages 1, 2, and 3 according to Hoehn and Yahr Classification

Exclusion Criteria:

* Severe cognitive impairment defined as ≤ 20 in Montreal Cognitive Assessment
* Score greater than or equal to 6 on the geriatric depression scale
* Severe respiratory and / or cardiovascular conditions
* Visual and / or auditory deficit that cannot be corrected with glasses or a hearing aid;
* Other previously detected orthopedic or neurological diseases, other than Parkinson's Disease, that may interfere with the individual's performance
* Previous experience with Microsoft XBOX Kinect® games
* And being in rehabilitation in another location concomitant to this training.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Balance Evaluation Systems Test (BESTest) | Change from baseline up to 3 months
  Balance Evaluation Systems Test (BESTest) measures balance. It includes 36 items that evaluate performance of 6 balance systems: biomechanical constraints, stability limits/verticality, anticipatory postural adjustments, postural responses, sensory orientation, and stability in gait.
International Falls Effectiveness Scale (FES-I) | Change from baseline up to 3 months
  It presents questions about the concern with the possibility of falling when performing 16 activities, with respective scores from one to four. The total score can range from 16 (no concern) to 64 (extreme worry).
30-second Gait Test | Change from baseline up to 3 months
  Functional mobility test that assesses gait performance under the influence of a verbal fluency cognitive task (speaking as many words that start with a certain letter established by the evaluator), in which the individual must walk continuously for 30 seconds and, when multitasking, he or she is instructed to perform both without interruption (command = "perform both tasks at the same time, without stopping talking or walking"). The evaluator measures the distance that the subject was able to travel in a single task and in a double task.
Six Minute Walk Distance | Change from baseline up to 3 months
  A gait assessment method that measures the maximum distance a person can walk in six minutes and measures maximal cardiorespiratory functions.
Five Times Sit to Stand | Change from baseline up to 3 months
  A measure of functional mobility that assists in the identification of insufficient strength and muscle strength of the lower limbs, assessing balance and identifying people at risk of falls. In this task, the individual is instructed to sit and get up from a chair, without armrests, for 5 times without stopping as quickly as possible. The evaluator measures the time the subject performs this task.
Unified Parkinson Disease Rating Scale - Session II | Change from baseline up to 3 months
  It is a gold standard scale used to assess and monitor PD progression. It consists of 42 items and divided into four segments: Part I (non-motor aspects of daily life), Part II (motor aspects of daily life), Part III (motor evaluation) and Part IV (motor complications). a score from 0 to 4 is established, the lower the score the better the individual's condition. In Part II, the questions are conducted by the evaluator and the answers are based on the self-reported report by the evaluated person regarding his motor performance in daily life activities.

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale - Session III | Change from baseline up to 3 months
  In session III of the UPDRS, the motor function is assessed, unlike session II which the score from 0 to 4 is given according to the individual's perception of his or her own performance, in this part the score is given according to the clinical motor analysis of the therapist. The higher the score, the worse the state of motor performance.
Rapid Turns Test | Change from baseline up to 3 months
  Measure of evaluation of the function related to the gait pattern, specifically to assess presence of episode of freezing of gait.
  The subject turns in a complete circle (360 degrees) as fast as he or she can while being timed to finish it. The test is done to both sides (right and left).
Geriatric Depression Scale | Change from baseline up to 3 months
  It is a test for detecting depressive symptoms in the elderly, with 15 questions in which the result of 5 or more points shows a sign of depression, with a score equal to or greater than 11 characterizing severe depression.
Montreal Cognitive Assessment | Change from baseline up to 3 months
  The instrument assesses different cognitive domains such as visuospatial and executive functions, naming, memory, attention, language, abstraction and orientation. The total score of the scale is 30 points and scores greater than or equal to 26 indicate normal performance.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PT, PhD, Study Director — University of Sao Paulo; Pâmela Y Igarasi Barbosa, PT, Principal Investigator — University of Sao Paulo; Amarilis Falconi, PT, Principal Investigator — University of Sao Paulo
Locations (1):
- Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy, School of Medicine, University of São Paulo, São Paulo, São Paulo, Brazil